CLINICAL TRIAL: NCT02039843
Title: Can Service Dogs Improve Activity and Quality of Life in Veterans With PTSD?
Acronym: SDPTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SDPTSD
Record Dates: First submitted 2014-01-07; First posted 2014-01-20 (Estimated); Results first posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-02

CONDITIONS: Post Traumatic Stress Disorders
Keywords: Post Traumatic Stress Disorder; Service Dog; Emotional Support Dog
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Emotional Support Dogs (Active Comparator): Participants paired with Emotional Support Dogs
  Emotional Support Dogs were required to pass the American Kennel Club Canine Good Citizen and the American Kennel Club Community Canine tests and be well-behaved and well-socialized.
  Interventions: Other: Emotional Support Dogs
- Service Dogs (Active Comparator): Participants paired with Service Dogs
  Service Dogs were required to pass the American Kennel Club Canine Good Citizen and the Assistance Dogs International Public Access tests and trained to complete five PTSD-specific tasks (lights, sweep, bring, block, & behind).
  Interventions: Other: Service Dogs

INTERVENTIONS:
Other: Emotional Support Dogs — Emotional Support Dogs were required to pass the American Kennel Club Canine Good Citizen and the American Kennel Club Community Canine tests and be well-behaved and well-socialized.
  Arms: Emotional Support Dogs
Other: Service Dogs — Service Dogs were required to pass the American Kennel Club Canine Good Citizen and the Assistance Dogs International Public Access tests and trained to complete five PTSD-specific tasks (lights, sweep, bring, block, & behind).
  Arms: Service Dogs

SUMMARY:
Service Dogs are trained to assist people with disabilities to accomplish tasks which permit the individual to be more functional in their home and social environment. Often the dogs are trained to help in the completion of activities of daily living and instrumental activities of daily living. Service Dogs are efficacious for individuals with disabilities, such as vision limitations, spinal cord injury and hearing problems. In addition, some mental health outcomes have improved with the introduction of a Service Dog. A research study was mandated in the Department of Defense Bill of 2010, to examine the efficacy of service dogs for Veterans with Post Traumatic Stress Disorder (PTSD). Together with the Cooperative Studies Program, the proponents have designed a research study to effectively meet the demands of the Bill and to provide timely research into an evolving field.

DETAILED DESCRIPTION:
Background: Service Dogs are trained to assist people with disabilities to accomplish tasks which permit the individual to be more functional in their home and social environment. Often the dogs are trained to help in the completion of activities of daily living and instrumental activities of daily living. Service Dogs are efficacious for individuals with disabilities, such as vision limitations, spinal cord injury and hearing problems. In addition, some mental health outcomes have improved with the introduction of a Service Dog. A research study was mandated in the Department of Defense Bill of 2010, to examine the efficacy of service dogs for Veterans with Post Traumatic Stress Disorder (PTSD). Together with the Cooperative Studies Program, the proponents have designed a research study to effectively meet the demands of the Bill and to provide timely research into an evolving field.

Study Primary Objective: To examine how limitations on activity and quality of life in Veterans with PTSD are impacted by the provision of a Service Dog versus an Emotional Support Dog.

Study Design: A prospective randomized study is proposed which has two randomized arms. Arm one of the study will be Veterans (n=110) randomized and paired with a Service Dog, which has been trained in 5 PTSD-specific tasks to assist with the Veteran's PTSD issues. Arm two (n=110) of the study will be Veterans randomized and paired with an Emotional Support Dog (a dog that provides support via emotional comfort). All Veterans, after confirmation of eligibility, will be randomized to receive a Service Dog or Emotional Support Dog and will be observed for a minimum of three months prior to receiving their dog. During this observation period, Veterans will be required to participate in a Dog Care Course to ensure they are aware of the demands dogs place on humans. Once a dog becomes available, the Veteran will be paired with a Service Dog or Emotional Support Dog. Pairing is the training process in which the Veteran is given instruction and practice in commanding and caring for their new service dog or emotional support dog. The pairing process for a service dog takes place at the contracted dog vendor's location; the pairing process for an emotional support dog takes place at the Veteran's home, facilitated by a VA Dog Trainer. Follow-up with the Veteran begins one week post pairing to track any dog behavior issues, and will continue after pairing for 18 months. Primary outcomes to be examined include limitations on Veteran activity (as measured by the WHO-DAS 2.0) and quality of life (measured by the VR-12). Secondary outcomes include PTSD symptoms (measured by the PCL-5), suicidal ideation (C-SSRS); depression (PHQ-9) and Sleep (PSQI). In addition, health care utilization, anger management (DAR), employment, and work productivity will also be examined. Study outcomes are assessed at baseline (prior to randomization), and at 3-month intervals after a Veteran is paired with a dog until 18 months post pairing. This multi-site study will be conducted at three locations nationwide.

ELIGIBILITY:
Inclusion Criteria:

1. Males and Females greater than> 18 years of age.
2. Referral from Mental Health provider that documents PTSD.
3. PTSD as a result of any trauma as determined by meeting DSM 5 diagnostic criteria.
4. Enrolled in mental health services at VA and has attended at least one visit in the 90 days prior to consent.

   * If individual not currently enrolled in mental health treatment decides to enroll in such then he/she may become eligible to participate in the study.
   * If individual enrolled in mental health treatment schedules and attends a mental health visit then he/she may become eligible to participate in the study.
5. Agrees to remain in mental health treatment throughout the duration of the study
6. Can adequately care for a dog .

   * Adequately caring for a dog requires that participants will be responsible for and able to provide food, water, protection, shelter, exercise, transportation, and treatment related to their assigned dog.
   * Adequately handling the dog means having the ability to give and reinforce obedience commands and control the dog using a leash.
7. Home environment is suitable for a dog.

   * If the home environment can be remedied the potential participant may become eligible to participate in the study.
   * If a participant moves home while enrolled in the study the new home must be suitable for a dog.
8. Home environment is structurally and geographically accessible to study staff.

   * If the home is geographically inaccessible to study staff and, the individual cannot remedy the situation unless he/she moves home. The study team will not encourage this. If a move takes place, it will be the individual's responsibility to re-contact the study team.
   * If the individual changes home residence while enrolled in the study, the new home must be geographically accessible to study staff. If it is inaccessible, the dog will be removed and the individual will be withdrawn from the study.
9. Is willing to accept randomization outcome.
10. Has someone to care for dog during extended absence of the participant.

    * If no one is available to care for the dog but the situation changes then the participant may become eligible to participate.
11. Others in home are agreeable to having dog.

    * If others in the home are not agreeable but at a later date the situation changes, then the potential participant may become eligible to participate.
12. Is willing and able to travel (by air or car) to training site for pairing.

    * If potential participant's unwillingness to travel to a training site changes, he/she may become eligible to participate. In this instance, it will be the individual's responsibility to re-contact the study team.
13. Individual has no household pets that would threaten the bonding and obedience training of an assigned study dog.

    * If a household dog lives inside the home and the home is partitioned such that there are two or more separate living spaces served by independent entrance/exits, and the individual does not live in a partition with a dog, then the individual can be eligible. If a household dog lives primarily outside the home in a rural area and the individual is not primarily responsible for feeding the dog on a daily basis, then the individual can be eligible.
    * If an individual has pets other than dogs that could interfere with bonding, the individual will be scheduled for the screening visits and the relationship will be assessed by the dog trainer.
    * If an individual has a household dog or other pet that prevents participation in the study but the situation changes, the individual may become eligible to participate. In this instance, it will be the individual's responsibility to re-contact the study team.
14. Individual can verbalize understanding of consent form, is willing to provide written informed consent and to follow study procedures.

Exclusion Criteria:

1. Hospitalization for mental health reasons in the past 6 months.

   * Once six months since hospitalization have passed, the individual may become eligible to participate in the study.
2. Aggressive behavior that would make it unsafe for dog.
3. Diagnosis of psychosis, delusions, dementia, moderate or severe alcohol/substance disorder (SUD), or moderate to severe traumatic brain injury as determined by the presence or absence of a condition following scoring of MINI responses or as documented in chart notes.

   SUD assessment (alcohol/non-alcohol):
   * Ineligibility is based on the presence of a Moderate (4-5 symptoms) to Severe (6+ symptoms) SUD as identified by the MINI within the previous 12-month period starting from date of the study MINI screening.
   * If a Moderate to Severe SUD has been documented or communicated by the referring clinician or potential participant, or is noted in the EMR prior to the initial MINI screening visit, individuals should be scheduled for their initial screening visit on a timeline commensurate with meeting the 12-month SUDs eligibility window.
   * If an individual is identified as ineligible during the initial screening visit (i.e. MINI SUDs score ≥4) he/she may be re-evaluated later at the discretion of the study team. Re-evaluations should be scheduled based on a timeline commensurate with meeting the 12-month SUDs eligibility window (absence of a Moderate to Severe SUD for the previous 12 months). If at re-evaluation the individual has <4 symptoms, he/she may become eligible to participate in the study.
4. Active suicidal intent as determined by a CPRS flag for suicidal intent or an endorsement of yes to question 5 (active suicidal ideation with specific plan and intent) on the C-SSRS completed at the Clinic Qualifying Visit.

   * An endorsement of yes to question 4 (Active Suicidal Ideation with Some Intent to Act, without Specific Plan) without endorsement of question 5 indicates that the individual needs additional assessment to determine eligibility.
5. Homicidal intent or cognitive disabilities that would preclude safety of dog and/or ability to participate in the study.
6. Social, mental or physical condition that prevents the potential participant from either giving informed consent or participating in the study.
7. Participation in another unapproved research trial.

   * If the individual is in another unrelated study and both the study Chair/PI of this and the other study consider participation in both studies to be acceptable then the individual may become eligible to participate in this study.
   * If the study Chair/PI of this and/or the other study consider participation in both studies to be unacceptable then, once participation in the other study is complete, the participant may become eligible to participate in this study. At that time, it will be the individual's responsibility to re-contact the study team.
8. Has chart note flag for violent/disruptive behavior.
9. Potential participants who are pregnant/who have a partner who is pregnant, or who currently have one or more children younger than age 5 in the household for more than 8 hours per day, one day a week will be excluded from the study.

   * If a participant or anyone else in the household becomes pregnant during the observation period, the participant will be excluded from the study.
   * Participants who have children in their home/become pregnant after being paired with a dog will be evaluated on a case-by-case basis (see Safety Monitoring of Children in the Home below).
   * After a total of 10 dogs have been placed with participants who have children between the ages of 5 and 10 years, and after each pairing has successfully reached and passed the 2-month home visit, this exclusion criterion will be revisited for potential inclusion of participants with children younger than 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2014-12-15 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joan Richerson, DVM, Study Chair — Tennessee Valley Healthcare System Nashville Campus, Nashville, TN
Locations (4):
- United States (4):
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - Iowa City VA Health Care System, Iowa City, IA, Iowa City, Iowa
  - VA Portland Health Care System, Portland, OR, Portland, Oregon
  - Tennessee Valley Healthcare System Nashville Campus, Nashville, TN, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Saunders GH, Biswas K, Serpi T, McGovern S, Groer S, Stock EM, Magruder KM, Storzbach D, Skelton K, Abrams T, McCranie M, Richerson J, Dorn PA, Huang GD, Fallon MT. Design and challenges for a randomized, multi-site clinical trial comparing the use of service dogs and emotional support dogs in Veterans with post-traumatic stress disorder (PTSD). Contemp Clin Trials. 2017 Nov;62:105-113. doi: 10.1016/j.cct.2017.08.017. Epub 2017 Aug 26. PMID 28844986

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Sixty participants of 287 consented participants were found to be ineligible for study randomization per study inclusion/exclusion criteria, resulting in 227 participants randomized.
Groups:
- Emotional Support Dog: Participants with Emotional Support Dogs
  Emotional Support Dogs were required to pass the American Kennel Club Canine Good Citizen and the American Kennel Club Community Canine tests and be well-behaved and well-socialized.
- Service Dogs: Participants with Service Dogs
  Service Dogs were required to pass the American Kennel Club Canine Good Citizen and the Assistance Dogs International Public Access tests and trained to complete five PTSD-specific tasks (lights, sweep, bring, block, & behind).
Period: Randomization and Observation Period
Arm/Group | Emotional Support Dog | Service Dogs
Started (Number of participants randomized to each arm.) | 113 | 114
Completed (Randomized participants paired with a study dog.) | 84 | 97
Not Completed | 29 | 17
Not completed — Adverse Event | 2 | 0
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 2 | 3
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Other reasons not paired with a study dog | 22 | 11
Period: Pairing With a Study Dog
Arm/Group | Emotional Support Dog | Service Dogs
Started | 84 | 97
Completed | 65 | 88
Not Completed | 19 | 9
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 1 | 4
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Other reasons for not completing study | 13 | 4

BASELINE CHARACTERISTICS:
Population: Randomized participants paired with a study dog.
Groups:
- Emotional Support Dog: Participants paired with Emotional Support Dogs
  Emotional Support Dogs were required to pass the American Kennel Club Canine Good Citizen and the American Kennel Club Community Canine tests and be well-behaved and well-socialized.
- Total: Total of all reporting groups
Arm/Group | Emotional Support Dog | Service Dogs | Total
Number analyzed (Participants) | 84 | 97 | 181
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.2 (13.25) | 51.8 (13.87) | 50.6 (13.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 22 | 36
  Male | 70 | 75 | 145
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 4 | 12
  Not Hispanic or Latino | 74 | 91 | 165
  Unknown or Not Reported | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 12 | 10 | 22
  White | 52 | 68 | 120
  More than one race | 15 | 16 | 31
  Unknown or Not Reported | 1 | 1 | 2
World Health Organization Disability Assessment Scale II (WHO-DAS 2.0) [Mean (Standard Deviation); unit: units on a scale] — The World Health Organization Disability Assessment Scale II (WHO-DAS 2.0) is a standardized measure for assessing health and disability levels. For the WHO-DAS 2.0 36-item, self-administered questionnaire, participants rate the difficulty they experience with each item on a 5-item scale: 'None,' 'Mild,' 'Moderate,' 'Severe' or 'Extreme/cannot do.' Standardized total disability scores ranging from 0 (no disability) to 100 (full disability) are obtained (WHO-DAS 2.0 manual, 2012). Population: The number analyzed is different from the analysis population due to one participant missing an assessment.
  units on a scale
    number analyzed (Participants) | 83 | 97 | 180
    (all) | 38.31 (16.23) | 35.78 (16.72) | 36.95 (16.50)
Veterans Rand 12-Item Health Survey - Physical Component Score (VR-12 PCS) [Mean (Standard Deviation); unit: T-score] — The Veterans Rand 12-Item Health Survey (VR-12) assesses health-related quality of life and includes a physical component score (PCS) assessing general health, physical functioning, role limitations, and bodily pain (Selim et al., 2009). The PCS score is standardized using a T-score transformation with a mean of 50 (which indicates the population mean) and a standard deviation (SD) of 10 to represent the population norm based on U.S. population in 1990. T-scores below 50 represent worse quality of life compared to the U.S. population norm, and those above 50 indicate better quality of life. Population: The number analyzed is different from the analysis population due to one participant missing an assessment at baseline.
  T-score
    number analyzed (Participants) | 83 | 97 | 180
    (all) | 40.16 (9.94) | 43.07 (11.20) | 41.73 (10.71)
Veterans Rand 12-Item Health Survey - Mental Component Score (VR-12 MCS) [Mean (Standard Deviation); unit: T-score] — The Veterans Rand 12-Item Health Survey (VR-12) assesses health-related quality of life and includes a mental component score (MCS) assessing emotional, vitality/mental health and social functioning (Selim et al., 2009). The MCS score is standardized using a T-score transformation with a mean of 50 (which indicates the population mean) and a standard deviation (SD) of 10 to represent the population norm based on U.S. population in 1990. T-scores below 50 represent worse quality of life compared to the U.S. population norm, and those above 50 indicate better quality of life. Population: The number analyzed is different from the analysis population due to one participant missing an assessment at baseline.
  T-score
    number analyzed (Participants) | 83 | 97 | 180
    (all) | 31.11 (10.62) | 30.68 (10.37) | 30.88 (10.46)

OUTCOME MEASURES:

1. Primary Outcome: World Health Organization Disability Assessment Scale II (WHO-DAS 2.0) Total Score
Description: The World Health Organization Disability Assessment Scale II (WHO-DAS 2.0) is a standardized measure for assessing health and disability levels. For the WHO-DAS 2.0 36-item, self-administered questionnaire, participants rate the difficulty they experience with each item on a 5-item scale: 'None,' 'Mild,' 'Moderate,' 'Severe' or 'Extreme/cannot do.' Standardized total disability scores ranging from 0 (no disability) to 100 (full disability) are obtained (WHO-DAS 2.0 manual, 2012).
Time Frame: Baseline and every 3 months after dog pairing up to 18 months post-pairing
Population: Participants randomized and paired with an emotional support dog or a service dog. The number of participants analyzed at each 3-month follow-up time point represents the number of individuals still participating in the study at that time point and completing the assessment. As this was a longitudinal study, attrition was expected and seen over time. Reasons for attrition are noted in the Participant Flow section under the 'Pairing With a Study Dog' Period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Emotional Support Dogs | Service Dogs
Number analyzed (Participants) | 84 | 97
score on a scale
  Baseline: number analyzed (Participants) | 83 | 97
  Baseline | 38.31 (16.23) | 35.78 (16.72)
  Month 3: number analyzed (Participants) | 76 | 95
  Month 3 | 41.76 (16.89) | 38.76 (16.46)
  Month 6: number analyzed (Participants) | 73 | 94
  Month 6 | 41.70 (17.62) | 36.73 (16.33)
  Month 9: number analyzed (Participants) | 70 | 92
  Month 9 | 43.07 (18.74) | 36.90 (17.29)
  Month 12: number analyzed (Participants) | 68 | 90
  Month 12 | 40.79 (17.36) | 36.76 (17.23)
  Month 15: number analyzed (Participants) | 66 | 88
  Month 15 | 43.48 (17.83) | 36.16 (17.69)
  Month 18: number analyzed (Participants) | 65 | 88
  Month 18 | 38.05 (17.79) | 33.43 (17.38)
Statistical Analysis 1: Comparison: Emotional Support Dogs vs Service Dogs; Test type: Superiority; p = 0.052, Mixed Models Analysis — Two-sided a priori alpha level was 0.05; Linear mixed repeated measures analysis on group difference in WHO-DAS score adjusted for gender, site, baseline score, time & timeXgroup interaction

2. Primary Outcome: Veterans Rand 12-Item Health Survey (VR-12): Physical Component Score (PCS)
Description: The 12-item, self-administered Veterans Rand 12-Item Health Survey (VR-12) assesses health-related quality of life. Two sub-scores are derived: 1) a Physical Component Score (PCS) assessing general health, physical functioning, role limitations, and bodily pain; and 2) a Mental Component Score (MCS) assessing emotional, vitality/mental health and social functioning (Selim et al., 2009). The PCS score is standardized using a T-score transformation with a mean of 50 (which indicates the population mean) and a standard deviation (SD) of 10 to represent the population norm based on U.S. population in 1990. T-scores below 50 represent worse quality of life compared to the U.S. population norm, and those above 50 indicate better quality of life.
Time Frame: Baseline and every 3 months after dog pairing up to 18 months post-pairing
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Emotional Support Dog | Service Dogs
Number analyzed (Participants) | 84 | 97
T-score
  Baseline: number analyzed (Participants) | 83 | 97
  Baseline | 40.16 (9.94) | 43.07 (11.20)
  Month 3: number analyzed (Participants) | 75 | 94
  Month 3 | 37.14 (10.86) | 39.05 (11.08)
  Month 6: number analyzed (Participants) | 71 | 94
  Month 6 | 35.78 (10.83) | 39.80 (11.59)
  Month 9: number analyzed (Participants) | 69 | 89
  Month 9 | 35.35 (11.32) | 39.07 (11.65)
  Month 12: number analyzed (Participants) | 68 | 89
  Month 12 | 35.73 (12.52) | 38.89 (11.44)
  Month 15: number analyzed (Participants) | 66 | 87
  Month 15 | 35.78 (11.42) | 39.48 (11.43)
  Month 18: number analyzed (Participants) | 63 | 87
  Month 18 | 37.30 (11.60) | 38.52 (11.71)
Statistical Analysis 1: Comparison: Emotional Support Dog vs Service Dogs; Test type: Superiority; p = 0.421, Mixed Models Analysis — 2-sided a priori alpha level was 0.05; Linear mixed repeated measures analysis on group difference in PCS score adjusted for gender, site, baseline score, time, and timeXgroup

3. Primary Outcome: Veterans Rand 12-Item Health Survey (VR-12): Mental Component Score (MCS)
Description: The 12-item, self-administered Veterans Rand 12-Item Health Survey (VR-12) assesses health-related quality of life. Two sub-scores are derived: 1) a Physical Component Score (PCS) assessing general health, physical functioning, role limitations, and bodily pain; and 2) a Mental Component Score (MCS) assessing emotional, vitality/mental health and social functioning (Selim et al., 2009). The MCS score is standardized using a T-score transformation with a mean of 50 (which indicates the population mean) and a standard deviation (SD) of 10 to represent the population norm based on U.S. population in 1990. T-scores below 50 represent worse quality of life compared to the U.S. population norm, and those above 50 indicate better quality of life.
Time Frame: Baseline and every 3 months after dog pairing up to 18 months post-pairing
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Emotional Support Dog | Service Dogs
Number analyzed (Participants) | 84 | 97
T-score
  Baseline: number analyzed (Participants) | 83 | 97
  Baseline | 31.11 (10.62) | 30.68 (10.37)
  Month 3: number analyzed (Participants) | 75 | 94
  Month 3 | 35.59 (10.32) | 35.81 (9.07)
  Month 6: number analyzed (Participants) | 71 | 94
  Month 6 | 36.71 (11.30) | 35.71 (8.91)
  Month 9: number analyzed (Participants) | 69 | 89
  Month 9 | 34.53 (10.59) | 36.39 (9.92)
  Month 12: number analyzed (Participants) | 68 | 89
  Month 12 | 37.32 (10.66) | 36.98 (10.83)
  Month 15: number analyzed (Participants) | 66 | 87
  Month 15 | 36.42 (10.15) | 37.72 (11.40)
  Month 18: number analyzed (Participants) | 63 | 87
  Month 18 | 39.04 (12.35) | 40.28 (9.33)
Statistical Analysis 1: Comparison: Emotional Support Dog vs Service Dogs; Test type: Superiority; p = 0.606, Mixed Models Analysis — 2-sided a priori alpha level was 0.05; Linear mixed repeated measures analysis on group difference in MCS score adjusted for gender, site, baseline score, time, and timeXgroup

4. Secondary Outcome: Pittsburgh Sleep Quality Index (PSQI) Global Score
Description: The Pittsburgh Sleep Quality Index (PSQI) is a self-administered survey used to assess sleep-related problems during the past month (Buysse, et al., 1989). The 19 items completed by the participant are grouped into seven components: (1) Sleep quality, (2) Sleep latency, (3) Sleep duration, (4) Habitual sleep efficiency, (5) Sleep disturbances, (6) Use of sleep medication, and (7) Daytime dysfunction. Each of the seven components are weighted equally on a 0-3 scale with 0 (better) to 3 (worse). These are summed to yield a global score with a range of 0-21 with higher scores indicating worse sleep quality.
Time Frame: Baseline and every 3 months after dog pairing up to 18 months post-pairing
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Emotional Support Dog | Service Dogs
Number analyzed (Participants) | 84 | 97
score on a scale
  Baseline: number analyzed (Participants) | 84 | 96
  Baseline | 14.26 (4.09) | 13.60 (3.85)
  Month 3: number analyzed (Participants) | 75 | 95
  Month 3 | 13.60 (4.79) | 12.51 (4.24)
  Month 6: number analyzed (Participants) | 73 | 94
  Month 6 | 13.10 (4.60) | 12.17 (4.13)
  Month 9: number analyzed (Participants) | 69 | 91
  Month 9 | 13.29 (4.59) | 12.36 (4.37)
  Month 12: number analyzed (Participants) | 68 | 90
  Month 12 | 13.24 (4.88) | 12.27 (4.34)
  Month 15: number analyzed (Participants) | 64 | 88
  Month 15 | 12.91 (4.64) | 12.02 (4.50)
  Month 18: number analyzed (Participants) | 65 | 87
  Month 18 | 12.54 (4.85) | 11.74 (4.33)
Statistical Analysis 1: Comparison: Emotional Support Dog vs Service Dogs; Test type: Superiority; p = 0.210, Mixed Models Analysis — 2-sided a priori alpha level was 0.05; Linear mixed repeated measures analysis on group difference in PSQI score adjusted for gender, site, baseline score, time, and timeXgroup

5. Secondary Outcome: Post-Traumatic Stress Disorder (PTSD) Civilian Checklist 5 (PCL-5) Score
Description: The Post-Traumatic Stress Disorder (PTSD) Civilian Checklist 5 (PCL-5) is a 20-item self-report measure that assesses the 20 Diagnostic and Statistical Manual of Mental Disorder, 5th edition (DSM-5) symptoms of PTSD. Each symptom is scored on a scale of 0 (not at all) through 4 (extreme). A total symptom severity score is calculated by summing the scores for each of the 20 items. Scores can range from 0 to 80 with higher scores representing greater PTSD symptom severity.
Time Frame: Baseline and every 3 months after dog pairing up to 18 months post-pairing
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Emotional Support Dog | Service Dogs
Number analyzed (Participants) | 84 | 97
score on a scale
  Baseline | 46.98 (14.70) | 48.33 (15.66)
  Month 3: number analyzed (Participants) | 76 | 95
  Month 3 | 41.96 (15.45) | 41.54 (15.14)
  Month 6: number analyzed (Participants) | 73 | 94
  Month 6 | 39.66 (16.43) | 39.39 (14.87)
  Month 9: number analyzed (Participants) | 70 | 92
  Month 9 | 41.04 (15.49) | 38.29 (15.04)
  Month 12: number analyzed (Participants) | 68 | 90
  Month 12 | 40.01 (17.60) | 35.48 (15.39)
  Month 15: number analyzed (Participants) | 66 | 89
  Month 15 | 41.23 (16.50) | 35.75 (16.18)
  Month 18: number analyzed (Participants) | 65 | 88
  Month 18 | 35.25 (17.00) | 31.66 (14.61)
Statistical Analysis 1: Comparison: Emotional Support Dog vs Service Dogs; Test type: Superiority; p = 0.036, Mixed Models Analysis — 2-sided a priori alpha level was 0.05; Linear mixed repeated measures analysis on group difference in PCL-5 score adjusted for gender, site, baseline score, time, and timeXgroup

6. Secondary Outcome: Patient Health Questionnaire (PHQ-9) Score
Description: The Patient Health Questionnaire (PHQ-9) assesses the severity of depression (Kroenke, et al., 2002). It consists of 9 depression symptom questions with response choices of 0 (not at all), 1 (several days), 2 (more than half of days), or 3 (nearly every day). The total score is calculated by adding together the symptom ratings for each of the 9 questions so that scores range from 0 to 27 (higher scores represent greater depression severity).
Time Frame: Baseline and every 3 months after dog pairing up to 18 months post-pairing
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Emotional Support Dog | Service Dogs
Number analyzed (Participants) | 84 | 97
score on a scale
  Baseline | 13.08 (5.94) | 12.79 (5.85)
  Month 3: number analyzed (Participants) | 76 | 95
  Month 3 | 11.46 (6.05) | 10.95 (5.47)
  Month 6: number analyzed (Participants) | 73 | 94
  Month 6 | 10.55 (6.03) | 10.03 (5.07)
  Month 9: number analyzed (Participants) | 70 | 92
  Month 9 | 11.53 (6.18) | 9.52 (4.80)
  Month 12: number analyzed (Participants) | 68 | 90
  Month 12 | 11.03 (6.31) | 9.97 (5.65)
  Month 15: number analyzed (Participants) | 66 | 88
  Month 15 | 11.47 (6.20) | 9.67 (5.79)
  Month 18: number analyzed (Participants) | 65 | 88
  Month 18 | 9.43 (6.24) | 8.19 (4.45)
Statistical Analysis 1: Comparison: Emotional Support Dog vs Service Dogs; Test type: Superiority; p = 0.079, Mixed Models Analysis — 2-sided a priori alpha level was 0.05; Linear mixed repeated measures analysis on group difference in PHQ-9 score adjusted for gender, site, baseline score, time, and timeXgroup

7. Secondary Outcome: Dimensions of Anger Reactions (DAR) Score
Description: The 7-item Dimensions of Anger Reactions (DAR) is a seven-item scale that assesses anger disposition directed to others (Forbes, et al.,2004). For each item, participants indicate the degree to which each statement describes their feelings and behavior on an 8-point scale ranging from 0 (not at all) to 8 (exactly so). Scores are totaled yielding a range of 0 to 56 with higher scores indicating greater anger disposition.
Time Frame: Baseline and every 3 months after dog pairing up to 18 months post-pairing
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Emotional Support Dog | Service Dogs
Number analyzed (Participants) | 84 | 97
score on a scale
  Baseline | 23.82 (14.64) | 21.85 (15.07)
  Month 3: number analyzed (Participants) | 76 | 95
  Month 3 | 23.21 (15.87) | 22.14 (14.28)
  Month 6: number analyzed (Participants) | 73 | 94
  Month 6 | 21.05 (16.32) | 20.35 (13.75)
  Month 9: number analyzed (Participants) | 70 | 92
  Month 9 | 23.97 (16.16) | 19.52 (13.22)
  Month 12: number analyzed (Participants) | 68 | 90
  Month 12 | 22.97 (15.57) | 18.58 (14.75)
  Month 15: number analyzed (Participants) | 66 | 89
  Month 15 | 22.32 (16.91) | 17.47 (14.24)
  Month 18: number analyzed (Participants) | 65 | 88
  Month 18 | 20.15 (16.63) | 15.90 (14.37)
Statistical Analysis 1: Comparison: Emotional Support Dog vs Service Dogs; Test type: Superiority; p = 0.155, Mixed Models Analysis — 2-sided a priori alpha level was 0.05; Linear mixed repeated measures analysis on group difference in DAR score adjusted for gender, site, baseline score, time, and timeXgroup

8. Secondary Outcome: Number of Participants Reporting Suicidal Behavior or Ideation (SBI) Derived From the Columbia Suicide Severity Rating Scale (C-SSRS)
Description: The Suicidal Behavior or Ideation (SBI) indicator derived from the Columbia Suicide Severity Rating Scale (C-SSRS) is dichotomized as the presence or absence of suicidal behavior or ideation. Presence of SBI is indicated by a "Yes" response to any one of the five suicidal behavior or the five suicidal ideation questions.
Time Frame: Baseline and every 3 months after dog pairing up to 18 months post-pairing
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Emotional Support Dog | Service Dogs
Number analyzed (Participants) | 84 | 97
Participants
  Baseline | 13 | 24
  Month 3: number analyzed (Participants) | 76 | 95
  Month 3 | 22 | 33
  Month 6: number analyzed (Participants) | 73 | 94
  Month 6 | 19 | 21
  Month 9: number analyzed (Participants) | 70 | 92
  Month 9 | 19 | 22
  Month 12: number analyzed (Participants) | 68 | 90
  Month 12 | 20 | 25
  Month 15: number analyzed (Participants) | 66 | 89
  Month 15 | 21 | 20
  Month 18: number analyzed (Participants) | 65 | 88
  Month 18 | 18 | 13
Statistical Analysis 1: Comparison: Emotional Support Dog vs Service Dogs; Test type: Superiority; p = 0.157, Mixed Models Analysis — 2-sided a priori alpha level was 0.05; Generalized linear mixed repeated measures analysis on group difference in SBI adjusted for gender, site, baseline SBI, time, and timeXgroup

9. Secondary Outcome: Number of Outpatient Visits to Non-Veterans Administration (VA) Healthcare Providers or Mental Health Providers
Description: Non-Veterans Administration (VA) healthcare utilization will be assessed using the "HERC non-VA utilization survey." This survey was created in 2011 by VA Health Economics Resource Center (HERC) investigators. The HERC non-VA utilization survey is self-administered and asks about outpatient and inpatient (including Emergency Room) visits to non-VA healthcare and/or non-VA mental health providers.
  Sample size (n) reflects the number of participants who provided self-reported non-VA healthcare use information at the time of data collection.
Time Frame: Baseline and every 3 months after dog pairing up to 18 months post-pairing
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of visits
Arm/Group | Emotional Support Dogs | Service Dogs
Number analyzed (Participants) | 84 | 97
number of visits
  Baseline: number analyzed (Participants) | 84 | 96
  Baseline | 1.6 (3.8) | 1.1 (4.8)
  Month 3: number analyzed (Participants) | 75 | 95
  Month 3 | 0.9 (2.6) | 0.5 (1.3)
  Month 6: number analyzed (Participants) | 73 | 94
  Month 6 | 1.0 (2.8) | 0.4 (1.4)
  Month 9: number analyzed (Participants) | 70 | 92
  Month 9 | 1.3 (3.5) | 0.5 (1.5)
  Month 12: number analyzed (Participants) | 68 | 90
  Month 12 | 0.9 (2.7) | 0.7 (2.5)
  Month 15: number analyzed (Participants) | 66 | 89
  Month 15 | 1.4 (3.3) | 0.5 (1.5)
  Month 18: number analyzed (Participants) | 65 | 88
  Month 18 | 0.9 (2.1) | 0.6 (1.8)
Statistical Analysis 1: Comparison: Emotional Support Dogs vs Service Dogs; Test type: Superiority; p = 0.430, Regression, Linear — p-value from random effects regression controlling for month and baseline outcome

10. Secondary Outcome: Number of Emergency Room Visits to Non-Veterans Administration (VA) Facilities
Description: as for outcome 9
Time Frame: Baseline and every 3 months after dog pairing up to 18 months post-pairing
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of visits
Arm/Group | Emotional Support Dogs | Service Dogs
Number analyzed (Participants) | 84 | 97
number of visits
  Baseline: number analyzed (Participants) | 83 | 96
  Baseline | 0.1 (0.4) | 0.1 (0.3)
  Month 3: number analyzed (Participants) | 75 | 95
  Month 3 | 0.1 (0.3) | 0.0 (0.2)
  Month 6: number analyzed (Participants) | 72 | 94
  Month 6 | 0.1 (0.3) | 0.0 (0.2)
  Month 9: number analyzed (Participants) | 70 | 92
  Month 9 | 0.1 (0.6) | 0.1 (0.3)
  Month 12: number analyzed (Participants) | 68 | 90
  Month 12 | 0.1 (0.4) | 0.1 (0.3)
  Month 15: number analyzed (Participants) | 66 | 89
  Month 15 | 0.1 (0.3) | 0.0 (0.2)
  Month 18: number analyzed (Participants) | 65 | 88
  Month 18 | 0.1 (0.3) | 0.1 (0.3)
Statistical Analysis 1: Comparison: Emotional Support Dogs vs Service Dogs; Test type: Superiority; p = 0.358, Regression, Linear — p-value from random effects regression controlling for month and baseline outcome

11. Secondary Outcome: Percentage of Participants With a Non-VA Hospitalization
Description: as for outcome 9
Time Frame: Baseline and every 3 months after dog pairing up to 18 months post-pairing
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of participants
Arm/Group | Emotional Support Dogs | Service Dogs
Number analyzed (Participants) | 84 | 97
Percentage of participants
  Baseline: number analyzed (Participants) | 84 | 96
  Baseline | 0 (0) | 6 (24)
  Month 3: number analyzed (Participants) | 76 | 94
  Month 3 | 3 (16) | 5 (23)
  Month 6: number analyzed (Participants) | 73 | 94
  Month 6 | 5 (23) | 2 (15)
  Month 9: number analyzed (Participants) | 70 | 91
  Month 9 | 3 (17) | 8 (27)
  Month 12: number analyzed (Participants) | 67 | 90
  Month 12 | 3 (17) | 3 (18)
  Month 15: number analyzed (Participants) | 66 | 88
  Month 15 | 0 (0) | 1 (11)
  Month 18: number analyzed (Participants) | 64 | 88
  Month 18 | 0 (0) | 2 (15)
Statistical Analysis 1: Comparison: Emotional Support Dogs vs Service Dogs; Test type: Superiority; p = 0.39, Regression, Linear — p-value from random effects regression controlling for month and baseline outcome

12. Secondary Outcome: Number of Outpatient Visits to Veterans Administration (VA) Healthcare Providers or Mental Health Providers.
Description: Utilization of VA outpatient services, identified using VA administrative data. The investigators identified all VA utilization and cost data for the 540 days (i.e., 18 months) starting on the date of pairing for each participant and summarized the data into six 90-day periods.
Time Frame: 540 days starting on the pairing date; summarized into six 90-day periods
Population: Participants randomized and paired with an emotional support dog or a service dog.
Measure: Mean (Standard Deviation); unit: number of visits
Arm/Group | Emotional Support Dogs | Service Dogs
Number analyzed (Participants) | 84 | 97
number of visits
  Baseline (90 days prior to pairing) | 16.4 (9.1) | 15.2 (10.6)
  Days 1-90 | 15.1 (9.3) | 15.1 (11.3)
  Days 91-180 | 14.5 (9.1) | 15 (9.8)
  Days 181-270 | 14.5 (10.1) | 14.4 (11.2)
  Days 271-360 | 13.4 (8.5) | 13.4 (9.8)
  Days 361-450 | 14.2 (8.7) | 13.8 (10.5)
  Days 451-540 | 14.8 (10.7) | 13 (9.8)

13. Secondary Outcome: Number of Inpatient Admissions to Veterans Administration (VA) Healthcare Providers or Mental Health Providers
Description: Utilization of VA inpatient services, identified using VA administrative data. The investigators identified all VA utilization and cost data for the 540 days (i.e., 18 months) starting on the date of pairing for each participant and summarized the data into six 90-day periods.
Time Frame: 540 days starting on the pairing date; summarized into six 90-day periods
Population: Participants randomized and paired with an emotional support dog or a service dog
Measure: Mean (Standard Deviation); unit: Number of inpatient admissions
Arm/Group | Emotional Support Dogs | Service Dogs
Number analyzed (Participants) | 84 | 97
Number of inpatient admissions
  Baseline (90 days prior to pairing) | 0 (0.1) | 0.1 (0.3)
  Days 1-90 | 0 (0.1) | 0.1 (0.3)
  Days 91-180 | 0 (0.2) | 0 (0.2)
  Days 181-270 | 0 (0.3) | 0.1 (0.3)
  Days 271-360 | 0 (0.1) | 0 (0.2)
  Days 361-450 | 0.1 (0.3) | 0.1 (0.4)
  Days 451-540 | 0 (0.3) | 0 (0.1)

14. Secondary Outcome: Total Cost of Outpatient Visits to Veterans Administration (VA) Healthcare Providers or Mental Health Providers
Description: Cost of VA outpatient services, identified using VA administrative data. The investigators identified all VA utilization and cost data for the 540 days (i.e., 18 months) starting on the date of pairing for each participant and summarized the data into six 90-day periods.
Time Frame: 540 days starting on the pairing date; summarized into six 90-day periods
Population: Participants randomized and paired with an emotional support dog or a service dog
Measure: Mean (Standard Deviation); unit: U.S. dollars
Arm/Group | Emotional Support Dogs | Service Dogs
Number analyzed (Participants) | 84 | 97
U.S. dollars
  Baseline (90 days prior to pairing) | 4701.32 (4714.98) | 4496.76 (4547.64)
  Days 1-90 | 3997.82 (3433.71) | 4696.70 (4363.93)
  Days 91-180 | 3684.87 (3295.50) | 4579.89 (4833.31)
  Days 181-270 | 3869.49 (4358.85) | 4360.64 (4602.07)
  Days 271-360 | 3494.07 (3840.25) | 4025.24 (4438.57)
  Days 361-450 | 3762.58 (3886.48) | 4043.37 (4333.64)
  Days 451-540 | 3685.47 (4648.30) | 3449.97 (4099.49)

15. Secondary Outcome: Total Cost of Inpatient Admissions to Veterans Administration (VA) Healthcare Providers or Mental Health Providers
Description: Cost of VA inpatient services, identified using VA administrative data. The investigators identified all VA utilization and cost data for the 540 days (i.e., 18 months) starting on the date of pairing for each participant and summarized the data into six 90-day periods.
Time Frame: 540 days starting on the pairing date; summarized into six 90-day periods
Population: Participants randomized and paired with an emotional support dog or a service dog
Measure: Mean (Standard Deviation); unit: U.S. dollars
Arm/Group | Emotional Support Dogs | Service Dogs
Number analyzed (Participants) | 84 | 97
U.S. dollars
  Baseline (90 days prior to pairing) | 184.53 (1701.29) | 1341.99 (7621.15)
  Days 1-90 | 132.36 (1220.31) | 727.11 (3513.19)
  Days 91-180 | 803.92 (5758.11) | 567.10 (3690.03)
  Days 181-270 | 1182.46 (8807.28) | 1219.27 (8693.99)
  Days 271-360 | 70.04 (456.89) | 1403.54 (6648.71)
  Days 361-450 | 916.85 (5527.54) | 1174.82 (6770.73)
  Days (451-540) | 439.40 (2943.53) | 333.03 (2311.15)

16. Secondary Outcome: Total Cost of VA Healthcare (Inpatient and Outpatient)
Description: Cost of VA inpatient and outpatient services, identified using VA administrative data. The investigators identified all VA utilization and cost data for the 540 days (i.e., 18 months) starting on the date of pairing for each participant and summarized the data into six 90-day periods.
Time Frame: 540 days starting on the pairing date; summarized into six 90-day periods
Population: Participants randomized and paired with an emotional support dog or a service dog
Measure: Mean (Standard Deviation); unit: U.S. dollars
Arm/Group | Emotional Support Dogs | Service Dogs
Number analyzed (Participants) | 84 | 97
U.S. dollars
  Baseline (90 days prior to pairing) | 4885.85 (5043.26) | 5838.74 (9613.11)
  Days 1-90 | 4130.18 (3637.66) | 5423.80 (6612.74)
  Days 91-180 | 4488.79 (7642.83) | 5146.99 (7084.47)
  Days 181-270 | 5051.95 (10019.56) | 5579.91 (9864.29)
  Days 271-360 | 3564.11 (3895.45) | 5428.78 (8514.41)
  Days 361-450 | 4679.42 (7081.99) | 5218.19 (8398.77)
  Days 451-540 | 4124.87 (6196.64) | 3782.99 (4929.90)

17. Secondary Outcome: Percentage of Days Covered for Antidepressants
Description: The investigators calculated Proportion of Days Covered (PDC) to measure medication adherence for common psychiatric medications dispensed by VA. Using the VA Drug Class variable, the investigators categorized medications into four categories: antidepressants (CN600-CN699), antipsychotics (CN700-CN799), benzodiazepine (CN302), and other hypnotics and sedatives (CN300, CN301, CN309). PDC for antidepressants are reported for this outcome (as a percentage).
Time Frame: Baseline: The 540 days prior to pairing Follow up: Pairing through day 540
Population: Participants with at least one refill in the drug class randomized and paired with an emotional support dog or a service dog
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | Emotional Support Dogs | Service Dogs
Number analyzed (Participants) | 84 | 97
Percentage of days
  Baseline: number analyzed (Participants) | 72 | 83
  Baseline | 78.10 (21.60) | 73.90 (23.20)
  Follow up: number analyzed (Participants) | 68 | 78
  Follow up | 70.50 (20.80) | 77.20 (21.80)

18. Secondary Outcome: Percentage of Days Covered for Antipsychotics
Description: The investigators calculated Proportion of Days Covered (PDC) to measure medication adherence for common psychiatric medications dispensed by VA. Using the VA Drug Class variable, the investigators categorized medications into four categories: antidepressants (CN600-CN699), antipsychotics (CN700-CN799), benzodiazepine (CN302), and other hypnotics and sedatives (CN300, CN301, CN309). PDC for antipsychotics are reported for this outcome (as a percentage).
Time Frame: Baseline: The 540 days prior to pairing Follow up: Pairing through day 540
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | Emotional Support Dogs | Service Dogs
Number analyzed (Participants) | 84 | 97
Percentage of days
  Baseline: number analyzed (Participants) | 15 | 16
  Baseline | 79.00 (22.40) | 72.30 (20.90)
  Follow up: number analyzed (Participants) | 14 | 16
  Follow up | 71.40 (28.50) | 76.30 (17.40)

19. Secondary Outcome: Percentage of Days Covered for Benzodiazepines
Description: The investigators calculated Proportion of Days Covered (PDC) to measure medication adherence for common psychiatric medications dispensed by VA. Using the VA Drug Class variable, the investigators categorized medications into four categories: antidepressants (CN600-CN699), antipsychotics (CN700-CN799), benzodiazepine (CN302), and other hypnotics and sedatives (CN300, CN301, CN309). PDC for benzodiazepines are reported for this outcome (as a percentage).
Time Frame: Baseline: The 540 days prior to pairing Follow up: Pairing through day 540
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | Emotional Support Dogs | Service Dogs
Number analyzed (Participants) | 84 | 97
Percentage of days
  Baseline: number analyzed (Participants) | 22 | 14
  Baseline | 61.60 (25.60) | 72.60 (26.60)
  Follow up: number analyzed (Participants) | 21 | 15
  Follow up | 54.80 (28.30) | 60.10 (29.30)

20. Secondary Outcome: Percentage of Days Covered for Other Sedatives
Description: The investigators calculated Proportion of Days Covered (PDC) to measure medication adherence for common psychiatric medications dispensed by VA. Using the VA Drug Class variable, the investigators categorized medications into four categories: antidepressants (CN600-CN699), antipsychotics (CN700-CN799), benzodiazepine (CN302), and other hypnotics and sedatives (CN300, CN301, CN309). PDC for other sedatives are reported for this outcome (as a percentage).
Time Frame: Baseline: The 540 days prior to pairing Follow up: Pairing through day 540
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | Emotional Support Dogs | Service Dogs
Number analyzed (Participants) | 84 | 97
Percentage of days
  Baseline: number analyzed (Participants) | 17 | 19
  Baseline | 66.90 (30.90) | 63.20 (25.30)
  Follow up: number analyzed (Participants) | 13 | 17
  Follow up | 79.10 (27.80) | 63.00 (21.50)

21. Secondary Outcome: Number of Veterans Employed
Description: Employment assessed using the question "Are you currently employed (working for pay)?" from the Work Productivity and Activity Impairment Questionnaire: General Health Problem V2.0 (WPAI V2.0; Reilly et al, 1993). Sample size (n) reflects the number of participants who provided work productivity and employment information at the time of data collection.
Time Frame: Baseline and every 3 months after dog pairing up to 18 months post-pairing
Population: Participants randomized and paired with an emotional support dog or a service dog
Measure: Count of Participants; unit: Participants
Arm/Group | Emotional Support Dogs | Service Dogs
Number analyzed (Participants) | 84 | 97
Participants
  Baseline | 28 | 25
  Month 3: number analyzed (Participants) | 76 | 95
  Month 3 | 27 | 22
  Month 6: number analyzed (Participants) | 73 | 94
  Month 6 | 23 | 23
  Month 9: number analyzed (Participants) | 70 | 92
  Month 9 | 20 | 22
  Month 12: number analyzed (Participants) | 68 | 90
  Month 12 | 19 | 21
  Month 15: number analyzed (Participants) | 66 | 89
  Month 15 | 18 | 25
  Month 18: number analyzed (Participants) | 65 | 88
  Month 18 | 17 | 21
Statistical Analysis 1: Comparison: Emotional Support Dogs vs Service Dogs; Test type: Superiority; p = 0.383, Regression, Linear — p-value from random effects regression controlling for month and baseline outcome

22. Secondary Outcome: Impact of Health on Work Productivity Score
Description: Impact of Health on Work Productivity was assessed using the Work Productivity and Activity Impairment Questionnaire: General Health Problem V2.0 (WPAI V2.0; Reilly et al, 1993). Only participants who were employed were included in this analysis. Scores can range from 0 (no impact of health on work productivity) to 10 (extreme impact of health on work productivity), so a higher score represents a greater impact of health on work productivity.
Time Frame: Baseline and every 3 months after dog pairing up to 18 months post-pairing
Population: Participants randomized and paired with an emotional support dog or a service dog
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Emotional Support Dogs | Service Dogs
Number analyzed (Participants) | 84 | 97
score on a scale
  Baseline: number analyzed (Participants) | 27 | 20
  Baseline | 5.7 (2.6) | 3.3 (2.2)
  Month 3: number analyzed (Participants) | 24 | 21
  Month 3 | 4.7 (2.6) | 3.4 (2.8)
  Month 6: number analyzed (Participants) | 21 | 22
  Month 6 | 4.1 (2.7) | 3.1 (2.9)
  Month 9: number analyzed (Participants) | 16 | 22
  Month 9 | 3.9 (2.9) | 2.7 (2.8)
  Month 12: number analyzed (Participants) | 17 | 21
  Month 12 | 3.1 (2.6) | 3.4 (2.6)
  Month 15: number analyzed (Participants) | 17 | 25
  Month 15 | 3.6 (2.2) | 3 (2.9)
  Month 18: number analyzed (Participants) | 15 | 19
  Month 18 | 2.7 (2.2) | 3.7 (2.3)
Statistical Analysis 1: Comparison: Emotional Support Dogs vs Service Dogs; Test type: Superiority; p = 0.932, Regression, Linear

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAE) were assessed continuously from the time of a participant's consent up to 19 months post-pairing (18 months post-pairing + 30 days). Other (non-SAE) adverse events were collected starting from dog pairing until up to 19 months post-pairing (18 months post-pairing + 30 days).
Description: For participants consented, all SAEs were collected. Other AEs were collected if possibly or definitely related to the intervention. Events AFTER pairing are reported under the randomized treatment group. Events BEFORE pairing are in the Prior to Dog Pairing group. Participants with an event in the Prior to Dog Pairing group may have an event reported in a treatment group. One SAE with a partial missing date is believed to have occurred prior to pairing and is in "Prior to Dog Pairing" group.
Groups:
- Emotional Support Dog: Participants randomized and paired to receive an Emotional Support Dog
  Emotional Support Dog - a dog that has earned AKC Good Canine Citizen certification and provides emotional support and comfort to the Veteran.
- Service Dog: Participants randomized and paired to receive a Service Dog
  Service Dog - an assistance dog specifically trained to perform tasks that are specific to the person's disability and has public access privileges.
- Prior to Dog Pairing: All participants consented regardless of whether eventually randomized and paired with a dog.
Arm/Group | Emotional Support Dog | Service Dog | Prior to Dog Pairing
All-Cause Mortality (participants affected / at risk) | 1/84 | 0/97 | 1/287
Serious Adverse Events (participants affected / at risk) | 21/84 | 18/97 | 18/287
Other Adverse Events (participants affected / at risk) | 5/84 | 0/97 | 1/287
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Emotional Support Dog (N=84) | Service Dog (N=97) | Prior to Dog Pairing (N=287)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (2) | 1 (1)
Coronary artery disease (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Postural orthostatic tachycardia syndrome (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0)
Prinzmetal angina (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis alcoholic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 2 (2) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (2) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infected skin ulcer (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 1 (2)
Post procedural infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cardiac procedure complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Heart rate decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (2)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 3 (4) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (3)
Alcoholism (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2)
Drug use disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Substance use disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 3 (3) | 6 (7) | 2 (2)
Suicide attempt (Psychiatric disorders) | 1 (1) | 1 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Social stay hospitalisation (Social circumstances) | 0 (0) | 1 (1) | 0 (0)
Alcohol detoxification (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Heart valve replacement (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0)
Liposuction (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Metabolic surgery (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Plastic surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Rehabilitation therapy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Spinal decompression (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Spinal operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Emotional Support Dog (N=84) | Service Dog (N=97) | Prior to Dog Pairing (N=287)
Allergy to animal (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Infestation (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Emotional distress (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-05-14): https://cdn.clinicaltrials.gov/large-docs/43/NCT02039843/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-15): https://cdn.clinicaltrials.gov/large-docs/43/NCT02039843/SAP_001.pdf